CLINICAL TRIAL: NCT02394691
Title: Effect of Daily Left Prefrontal Dorsolateral Transcranial Direct Current Stimulation Sessions on Cognitive Improvement in Patients With Disorders of Consciousness
Brief Title: Effect of Repeated tDCS Sessions on Cognitive Improvement in Patients With Disorders of Consciousness
Acronym: rtDCS in DOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Aurore Thibaut, MSc, University of Liege
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014/113
Record Dates: First submitted 2015-03-11; First posted 2015-03-20 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Disorders of Consciousness; Severe Brain Injury; Post-comatose Non-communicative Patients
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal stimulation (Active Comparator): Patients receive an anodal tDCS (on the left dorsolateral prefrontal cortex) every day for 4 weeks, 5 days per week (tDCS of 2mA during 20minutes). A CRS-R is performed at baseline (before the first stimulation) and after the tDCS session. A final CRS-R is performed 8 week after the end of the session to assess the potential long term effects of tDCS.
  Interventions: Device: transcranial direct current stimulation
- sham stimulation (Placebo Comparator): Patients receive a sham tDCS (on the left dorsolateral prefrontal cortex) every day for 4 weeks, 5 days per week (tDCS of 2mA during 5 secondes at the begining and the end of the stimulation to mimic the effects of tDCS). A CRS-R is performed at baseline (before the first stimulation) and after the tDCS session. A final CRS-R is performed 8 week after the end of the session to assess the potential long term effects of tDCS.
  Interventions: Device: transcranial direct current stimulation

INTERVENTIONS:
Device: transcranial direct current stimulation — anodal transcranial direct current stimulation on the left dorsolateral prefrontal cortex for the anodal session and sham stimulation (5secondes of tDCS) for the sham session

SUMMARY:
In this study, researchers will show to caregivers of patients how to use a tDCS device (this device was designed to be easy to use, with fixed parameters and only one button to press to run the stimulation). They will be asked to apply a stimulation every day, 5 days per week during for 4 weeks, in chronic patients in minimally conscious state (MCS).

2 sessions of 4 weeks of stimulations will be realized, one anodal and one sham in a randomized order. Before and after each session, behavioral improvement will be assessed with the Coma Recovery Scale Revised (CRS-R). A final assessment will be done 8 weeks after the end of the sessions to assess the long term effect of tDCS.

DETAILED DESCRIPTION:
A single session of tDCS showed positive effects on patients in MCS (study published in Neurology, 2014). Nevertheless, the effects went down after 1 or 2 hours. In a second study (Protocol ID: 2009/201/B) we have found that 5 days of tDCS increase the lasting of the effects up to one week.

To know if tDCS could be use in clinical daily practice, a new study will evaluate the effects of 20 minutes of tDCS over the left prefrontal dorsolateral cortex for 4 weeks, 5 days per week, in chronic patients in MCS.

2 sessions of 4 weeks of stimulation (total=20 stimulations per session) will be performed, one session will be real (anodal stimulation) and one placebo (sham stimulation).

Firstly, the patient will be seen at the hospital for a behavioral assessment (CRS-R) with one of his/her caregiver. The investigator will explain to the caregiver how to perform the stimulation. In addition, he/she will receive a folder and a video. The caregiver will take an exam to be sure he/she performs the tDCS properly.

Before and after each stimulation session, behavioral improvement will be assessed with the CRS-R by a trained neuropsychologist, at the hospital. A final assessment will be done 8 weeks after the end of the session to assess the long term effect of tDCS.

The compliance will be recorded by the deice to be sure that the caregiver performs the stimulation every day as expected.

Researchers expect to see (a) an improvement of the CRS-R total score at the end of the anodal session and (b) this improvement persists for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* be in an minimally conscious state
* be chronic (more then 3 months post insult)
* stable condition

Exclusion Criteria:

* NMDA receptor inhibitor drugs
* modification of the treatment during the protocol
* illness or infection during the protocol
* pacemaker
* metallic cerebral implant
* prior neurological disorder
* tDCS or other non-invasive brain stimulation treatment less than 3months before the inclusion in the present study

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in the CRS-R total score | after each stimulation sessions (4 weeks) and 8 weeks later
  Improvement of the CRS-R total score after the end of the anodal session and 8 weeks later but no change for the sham session.
Safety of the device (adverse effect) | Recorded after each stimulations sessions (4 weeks) and 8 weeks later
  a questionnaire will be asked to the caregivers and family of the patient to know any adverse effect (drowsiness, redness of the skin, epileptic sizure, sign of pain or discomfort).
Usability of the device in daily clinical practice (compliance of the device by the caregivers) | After the end of the protocol (24 weeks)
  The tDCS device records the number of stimulations performed during the protocol. We will be able to evaluate the compliance of the device by the caregivers to know if they use it properly and as expected.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Liège, Liège, Liège, Belgium

REFERENCES:
- [Result] Thibaut A, Bruno MA, Ledoux D, Demertzi A, Laureys S. tDCS in patients with disorders of consciousness: sham-controlled randomized double-blind study. Neurology. 2014 Apr 1;82(13):1112-8. doi: 10.1212/WNL.0000000000000260. Epub 2014 Feb 26. PMID 24574549